CLINICAL TRIAL: NCT06979479
Title: Effectiveness of the Adapt for Life, Mental Wellness and Suicide Prevention Program
Acronym: AFL
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Drew Barzman, MD, Director of the Child & Adolescent Forensic Research Program Director of Research for the UC Division of Forensic Psychiatry Professor of Psychiatry, Children's Hospital Medical Center, Cincinnati
Other Study IDs: 2019-1334
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Depression Disorders; Suicidality
Keywords: Mental Health; Wellbeing; Stress Management; ADAPT Framework
MeSH Terms: conditions — Suicidal Ideation; Psychological Well-Being | interventions — Acclimatization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: These participants took all three surveys before receiving the AFL 4-day course. They instead, were given the AFL 4-day course the following semester.
- Experimental: These participants took the baseline survey prior to the AFL 4-day course. They then participated in the AFL 4-day course. Immideately after, they took the post-test survey and a 3 month follow up test, 3 months post.
  Interventions: Behavioral: school-based intervention

INTERVENTIONS:
Behavioral: school-based intervention — AFL is a four-day program aimed at combating the stigma associated with mental health conditions and reducing suicidal ideation among youth. The program focuses on improving knowledge about depression and mental illness, enhancing self-efficacy skills for coping and seeking help, and increasing receptiveness to receiving assistance. Facilitated by mental health experts, the educational curriculum equips youth with the necessary tools to address feelings of hopelessness.
  Other Names: Adapt for Life
  Groups: Experimental

SUMMARY:
Adapt for Life is a mental health and wellbeing program designed to help young people develop healthy behaviors and important life skills to manage stress and mental health challenges. The program is a collaboration between Adapt for Life and Cincinnati Children's Hospital Medical Center.

Purpose of the Study: The primary purpose of the Adapt for Life study is to evaluate the effectiveness of the ADAPT framework in improving mental health outcomes for students. The framework includes steps such as Ask, Describe, Assess, Plan, and Talk, which are designed to help students tackle stress during everyday moments or in times of crisis.

Question the Study is Trying to Answer: The study seeks to answer whether the ADAPT framework can significantly improve students' ability to manage stress, recognize mental health issues, and seek appropriate help. It aims to determine if the program can reduce instances of harmful behaviors and improve overall mental wellbeing among participants.

DETAILED DESCRIPTION:
Purpose: The Adapt for Life study aims to evaluate the effectiveness of the ADAPT framework in improving mental health outcomes for students. The framework includes steps such as Ask, Describe, Assess, Plan, and Talk, which are designed to help students manage stress during everyday moments or in times of crisis.

Study Design: This study is a randomized controlled trial involving students from various schools in the Greater Cincinnati Tri-State area. Participants are randomly assigned to either the intervention group, which receives the ADAPT framework training, or the control group, which receives standard mental health education.

Intervention: The ADAPT framework consists of the following components:

Ask: Encouraging students to ask questions and seek help when needed. Describe: Helping students describe their feelings and experiences accurately. Assess: Teaching students to assess their mental health and stress levels. Plan: Guiding students in planning healthy coping strategies. Talk: Promoting open conversations about mental health. Hypothesis: The study hypothesizes that students who receive the ADAPT framework training will show significant improvements in their ability to manage stress, recognize mental health issues, and seek appropriate help compared to those who receive standard mental health education.

Outcome Measures: Primary outcomes include changes in students' self-reported stress levels, mental health awareness, and help-seeking behaviors. Secondary outcomes include reductions in harmful behaviors and improvements in overall mental wellbeing.

Data Collection: Data will be collected through REDCap surveys, interviews, and observational assessments conducted at baseline, post-intervention, and 3 month post-intervention stages.

Analysis: Statistical analyses will be performed to compare the outcomes between the intervention and control groups. Mixed-methods approaches will be used to assess the qualitative and quantitative aspects of the intervention's effectiveness.

Ethical Considerations: The study will adhere to ethical guidelines for research involving human subjects. Informed consent will be obtained from all participants and their guardians. Confidentiality and privacy will be maintained throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Student in 8th-12th grade

Exclusion Criteria:

* Non-English Speaking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Students from 12 high schools in the Greater Cincinnati area. The participants are 8th and 9th-grade students, with a total sample size of 1,102 records. The schools are demographically and socioeconomically paired, and health classes within each school are randomized into control and experimental groups.
Sampling Method: Probability Sample
Enrollment: 1102 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Improved self-efficacy | Enrollment - 3 Month Follow Up
  Improved Self-Efficacy:
  Definition: Self-efficacy is a student's belief in their ability to effectively manage stress and mental health challenges.
  Measurement: It is assessed through self-reported surveys where students rate their confidence in handling stressful situations and their ability to use coping strategies taught in the ADAPT framework.
  Survey Questions: Students answer questions about their perceived ability to manage anxiety, cope with academic pressure, and maintain emotional balance.
  Criteria: Higher scores on these surveys indicate greater self-efficacy, suggesting that students feel more capable of managing their mental health. This includes their confidence in applying techniques like mindfulness, problem-solving, and seeking support when needed.
  Impact: Improved self-efficacy can lead to better academic performance, healthier relationships, and overall enhanced wellbeing.
Improved Help-Seeking Attitudes | Enrollment - 3 Month Follow Up
  Improved Help-Seeking Attitudes:
  Definition: Help-seeking attitudes refer to a student's willingness to seek support from peers, educators, or mental health professionals when facing mental health challenges.
  Measurement: Evaluated through surveys and interviews where students express their likelihood of seeking help and their comfort level in discussing mental health issues.
  Survey Questions: Students answer questions about their willingness to talk to a teacher, counselor, or friend when feeling stressed or overwhelmed.
  Criteria: Positive changes are indicated by increased willingness to seek help and greater openness in discussing mental health concerns. Higher scores suggest students are more likely to reach out for support and feel comfortable sharing their struggles.
  Impact: Improved help-seeking attitudes can lead to earlier intervention, better mental health outcomes, and a supportive school environment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided